CLINICAL TRIAL: NCT04265287
Title: Severe Pneumonia In Children (S-PIC) Study: A Comparative Effectiveness Study Of Children With Severe Pneumonia In Asia
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore Clinical Research Institute (Other); Singhealth Foundation (Other Government)
Responsible Party: Principal Investigator, Jan Hau Lee, Senior Consultant, KK Women's and Children's Hospital
Other Study IDs: S-PIC
Record Dates: First submitted 2020-01-07; First posted 2020-02-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Pneumonia
Keywords: severe pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with severe pneumonia: Pediatric patients admitted to PICU due to severe pneumonia
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Demographic, clinical, microbiological, critical care support and management data will be collected.

SUMMARY:
Severe pneumonia is a leading cause of mortality and morbidity in children worldwide. Mortality rates from pediatric severe pneumonia are three times higher in South East Asia compared to the Western hemisphere. The lack of description of epidemiology, current management strategies and outcomes of children with severe pneumonia admitted to pediatric intensive care units (PICUs) in Asia is a barrier to improving pediatric critical care in the region. The lack of a sustainable pediatric critical care network in Asia makes multinational PICU studies challenging.

Through the Pediatric Acute & Critical Care Medicine Asian Network (PACCMAN), the investigators aim to estimate the burden of pediatric patients admitted to Asian PACCMAN PICUs due to severe pneumonia that develop pediatric acute respiratory distress syndrome. The investigators will characterize etiologies, identify risk factors associated with morbidity and mortality, and develop prognostic prediction models. The investigators hypothesize that there are non-modifiable (e.g., etiological agents) and modifiable risk factors (e.g., steroid therapy and ventilator strategies) that are associated with poor clinical outcomes.

To achieve these aims, the investigators propose a prospective multicenter cohort study over 24 months to recruit 2000 children with severe pneumonia. Pertinent demographic, clinical, microbiological, critical care support and management data will be collected to enable an investigation of the association between risk factors and clinical outcomes in these children. Upon completion of this large observational study, the investigators will have a rich database with detailed information on epidemiology, management strategies and clinical outcomes for severe pneumonia in Asian children.

DETAILED DESCRIPTION:
The Pediatric Acute & Critical Care Medicine Asian Network (PACCMAN) is the first pediatric critical care network in Asia. Through this network and this study, the investigators aim to provide a comprehensive epidemiological description, clinical management and outcomes of critically ill children with severe pneumonia across multiple sites in Asia. Through PACCMAN, the investigators aim to collect clinical data across at least 10 countries on children admitted to PICUs for severe pneumonia. Detailed data on aetiologies (not limited to vaccine-preventable pneumonia), broad age groups (not limited to a specific age group of children), and specific and supportive therapies in the PICU, will allow the investigators to perform comparative analysis of important non-modifiable and modifiable risk factors associated with mortality and functional outcomes in a large cohort of children with severe pneumonia. This sets the stage for multi-center studies to investigate the effectiveness of intensive care therapies on the outcomes of children with severe pneumonia.

The overall aim is to study the epidemiology of severe pneumonia is Asian children and compare the effectiveness of currently employed management strategies (related to invasive mechanical ventilation, adjunct and metabolic support) on clinical outcomes in approximately 2000 children with severe pneumonia admitted to PICUs across at least 10 countries in Asia.

The specific aims of this study are as follows:

Primary Aim: To (1) estimate the percentage of pediatric patients admitted to PACCMAN PICUs due to severe pneumonia; (2) estimate the percentage of pediatric patients admitted to PICUs for severe pneumonia that develop pediatric acute respiratory distress syndrome (PARDS) prior to PICU discharge or transfer; (3) estimate the overall and PARDS-specific mortality rates for children admitted for severe pneumonia; (4) characterize/classify etiologies of severe pneumonia according to the WHO criteria.

Secondary Aim 1: Obtain distributions and estimates of 28-day ventilation free days and 28-day PICU free days; estimate the proportion of patients requiring extracorporeal membrane oxygenation.

Secondary Aim 2: Identify risk factors associated with morbidity and mortality rates in children with severe pneumonia in Asia.

ELIGIBILITY:
Inclusion Criteria:

1. Children < 18 years old.
2. Admitted to one of the PICUs in the collaborative network.
3. Evidence of acute infection as defined as reported fever, documented fever or hypothermia, leukocytosis or leucopenia.
4. Evidence of acute respiratory illness as defined as new cough or sputum production, chest pain, dyspnea, tachypnea, abnormal respiratory examination findings or respiratory failure.
5. Radiological evidence of pneumonia within 72 hours before or after admission.

Exclusion Criteria:

1. Children with active do-not-resuscitate (DNR) orders
2. Children that have already been enrolled in this study within the previous 28 days
3. Have an alternative diagnosis of a respiratory disorder

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All PICU admission will be screened daily and those who meet the inclusion criteria will be recruited and consented (if necessary). The investigators will include all patients who are admitted to the PICU including those with oxygen therapy, non-invasive ventilation and invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 931 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of pediatric patients admitted to PACCMAN PICUs due to severe pneumonia | Throughout the study, over 24 months
  Estimate the percentage of pediatric patients admitted to PACCMAN PICUs due to severe pneumonia
Percentage of pediatric patients admitted to PICUs for severe pneumonia that develop pediatric acute respiratory distress syndrome (PARDS) prior to PICU discharge or transfer | Throughout the study, over 24 months
  Estimate the percentage of pediatric patients admitted to PICUs for severe pneumonia that develop pediatric acute respiratory distress syndrome (PARDS) prior to PICU discharge or transfer
Overall and PARDS-specific mortality rates for children admitted for severe pneumonia | Throughout the study, over 24 months
  Estimate the overall and PARDS-specific mortality rates for children admitted for severe pneumonia
Characterize/classify etiologies of severe pneumonia in children | Throughout study period, over 24 months
  Incidence of viral, bacterial and fungal severe pneumonia in children based on microbiological investigations performed as per standard of care.

SECONDARY OUTCOMES:
Obtain distributions and estimates of 28-day ventilation free days in patients with severe pneumonia. | Up to 28 days of mechanical ventilation
  Obtain distributions and estimates of 28-day ventilation free days.
Obtain distributions and estimates of 28-day PICU free days. | Up to 28 days of PICU stay
  Obtain distributions and estimates of 28-day PICU free days.
Estimate the proportion of patients severe pneumonia requiring extracorporeal membrane oxygenation. | Throughout the study period, 24 months
  Total number of patients and proportion of patients with severe pneumonia requiring extracorporeal membrane oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hau Lee, Principal Investigator — KK Women's and Children's Hospital, SingHealth
Locations (1):
- KK Women and Children Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Wong JJM, Abbas Q, Wang JQY, Xu W, Dang H, Phan PH, Guo L, Lee PC, Zhu X, Angurana SK, Pukdeetraipop M, Efar P, Yuliarto S, Choi I, Fan L, Hui AWF, Gan CS, Liu C, Samransamruajkit R, Cho HJ, Ong JSM, Lee JH; Pediatric Acute and Critical Care Asian Network (PACCMAN). Severe Pneumonia in PICU Admissions: The Pediatric Acute and Critical Care Medicine Asian Network (PACCMAN) Observational Cohort Study, 2020-2022. Pediatr Crit Care Med. 2024 Nov 1;25(11):1035-1044. doi: 10.1097/PCC.0000000000003598. Epub 2024 Aug 23. PMID 39177431